CLINICAL TRIAL: NCT01652222
Title: Experimental Study to Validate the "Therapeutic Game" CONEM-BETA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barcelonabeta Brain Research Center, Pasqual Maragall Foundation (Other)
Collaborators: Fundacion SARquavitae (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CONEM-BETA-FPM/SAR-0111
Record Dates: First submitted 2012-07-25; First posted 2012-07-27 (Estimated); Last update posted 2014-07-09 (Estimated); Status verified 2014-07

CONDITIONS: Alzheimer's Disease; Dementia
Keywords: Alzheimer; caregiver; dementia; social support; Montessori; Therapeutic game
MeSH Terms: conditions — Alzheimer Disease; Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- CONEM-BETA + socio-educational training (Experimental): Caregivers will receive 4 socioeducational training sessions during an 8 week period. These sessions will focus on the description and process of the Alzheimer's disease (AD), and will also provide to the caregivers resources and strategies to cope with AD. During the last 4 weeks, they will also systematically play with the patient at home with the CONEM-BETA game.
  After that period, caregivers will use the game based on their preference and frequence during a period of 6 more weeks.
  Interventions: Other: CONEM-BETA + socio-educational training
- Socio-educational training only (Active Comparator): Caregivers will receive the same 4 socioeducational training sessions as the experimental group, during an 8 week period.
  Interventions: Other: Socio-educational training only
- Control (No Intervention): Caregivers of this group will behave with his/her patient during the trial as they have been doing so far, but will receive no intervention

INTERVENTIONS:
Other: CONEM-BETA + socio-educational training — 4 socio-educative training sessions during 8 weeks, and caregivers will systematically play with their patients with CONEM-BETA therapeutic game during the last 4 weeks. The dyads will be assessed (primary timepoint). Caregivers will then continue using the game with their patients for an extra 6 weeks period as needed, to assess adherence and games preferences.
  Arms: CONEM-BETA + socio-educational training
Other: Socio-educational training only — 4 socio-educative training sessions during 8 weeks
  Arms: Socio-educational training only

SUMMARY:
The purpose of the study is to assess the efficacy of the systematic application of the CONEM-BETA game in the subjective welfare of family caregivers of patients with Alzheimer's disease or other advanced stage dementia.

DETAILED DESCRIPTION:
Alzheimer's disease (AD) is clinically diagnosed based on memory and cognitive deterioration, and the loss of other functional abilities. Nevertheless, for the caregivers and the patients themselves, the psychological and behavioral symptoms of dementia (PBSD) are specially relevant aspects.

These PBSD are a source of stress for the caregiver. PBSD treatment starts with non-pharmacological treatment, but if the symptomatology is moderate to severe, then pharmacological treatments are indicated on top of the non-pharmacological ones. The symptoms that better respond to non-pharmacological interventions are depression and mild apathy, wanderings and repetitive behaviors.

Once dementia progresses, the ability to interact at cognitive and emotional levels are reduced, and then, alternative approaches are needed. In this circumstance, it has been postulated that the caregivers should not try to bring -patients with AD back to the objective reality, but that they should rather empathize with them and establish an emotional connection. This is a complex process, and requires intervention tools that favor this connection and improve the subjective welfare of the caregivers of persons with dementia.

The current study is based on a previous experience in implementing the Montessori method at SARquavitae nursing homes and daycare centers. The "therapeutic game" called CONEM-BETA contains a subset of these activities that have been adapted from the original texts from the Myers Research Institute. We aim to prove that CONEM-BETA may have also socio-emotional benefits for the caregivers when they systematically use them at home with their AD relatives. These potential benefits will be assessed by using validated questionnaires that measure changes in subjective welfare, anxiety and depression, coping strategy, overload level and perceived social support.

ELIGIBILITY:
Inclusion Criteria Family Caregivers:

* to be a family caregiver of an person diagnosed with possible or probable Alzheimer's disease or other advanced stage dementia
* show interest in participating
* Sign informed consent

Inclusion Criteria Alzheimer's or dementia person:

* to have a probable or possible Alzheimer type dementia or other advanced dementia according to a diagnosis done by a Specialized Evaluation Unit
* GDS 5-6 and a minimental equal or lower than 12.
* to preserve a verbal comprehension of basic instructions
* to preserve the mobility of the arms, as well as the visual and auditive capacities that allow to conduct the activities.

Exclusion Criteria Caregivers:

* to have a negative attitude towards the emotional interaction with his/her Alzheimer or dementia family member
* Unavailability
* to participate in other socio-educative interventions during the study period.
* Any other situation that makes the caregiver as not suitable according to investigator's criteria

Exclusion Criteria Alzheimer's or dementia person:

* Do not have the sensorial or motor capacities needed for the interaction.
* Serious impairment of the verbal comprehension
* Disabling health conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2012-01; Primary Completion 2012-07 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
change from baseline compared to the control and active arms using the EBP questionnaire (subjective welfare of family caregivers of patients with possible or probable Alzheimer or other advanced stage dementia) | 8 weeks
  The EBP (Escala de Bienestar Psicologico - Psychological Welfare Scale) assesses the degree of the person self-satisfaction, comfort with himself during a period of his life, and contains four sub-scales: subjective welfare, material welfare, professional welfare and welfare of the relationship with his partner. It allows also to obtain partial scores, that allow to have indicators of overall welfare psychological index, and a weighted score obtained from the items with higher discriminative power

SECONDARY OUTCOMES:
change from baseline compared to the control and active arms using the Cornell scale and NPI-Q to assess behaviour of the patients with probable or possible Alzheimer's disease or other advanced stage dementia | 8 weeks
  Cornell scale assesses the signs associated with depressive disorders in patients with dementia. It contains 19 items that assess 5 dimensions of depression: changes in mood, behavior disorders, physical signs, circadian rhythms, and judgement disorders. NPI-Q is based on NPI (Neuropsychiatric Inventory), and was designed as screening tool to assess the emotional distress of the caregiver. NPI-Q assesses the degree of delusions, hallucinations, agitation, depression, anxiety, euphoria, apathy, disinhibition and irritability.
change from baseline compared to the control and active arms using the Martin and cols. scale to assess the overload level of the family caregivers of patients with probable or possible Alzheimer's disease or other advanced stage dementia | 8 weeks
  Martin and cols. scale is an adaptation of the Zarit questionnaire to assess the overload level of the caregiver. It is a self administered questionnaire, with 22 items.
change from baseline compared to the control and active arms using the Goldberg's scale to assess anxiety and depression of the family caregivers of patients with probable or possible Alzheimer's disease or other advanced stage dementia | 8 weeks
  The Goldberg's questionnaire has two subscales with 9 items each, one for anxiety and one for depression. It was originally designed by Goldberg with the aim of having a short interview as a screening tool.
change from baseline compared to the control and active arms using the DUKE-UNC scale to assess the perceived social support of the family caregivers of patients with probable or possible Alzheimer's disease or other advanced stage dementia | 8 weeks
  Developed for the general population, the DUKE-UNC questionnaire allows to assess the perceived social support. It is self-administered and contains 11 items.
change from baseline compared to the control and active arms using the PANAS scale to assess the changes in positive and negative affect of the caregivers of patients with probable or possible Alzheimer's disease or other advanced stage dementia | 8 weeks
  The PANAS questionnaire includes 20 items, 10 related to the impact on positive affect (PA), and 10 related to the negative impact in affect (NA).

CONTACTS AND LOCATIONS:
Overall Officials: Iciar Ancizu, PhD, Principal Investigator — SARquavitae, Barcelona, Spain; Sandra Poudevida, PhD, Principal Investigator — Pasqual Maragall Foundation, Barcelona, Spain
Locations (3):
- Spain (3):
  - Hospital de Santa Maria, Lleida, Catalonia
  - Hospital de Salt, Salt, Catalonia
  - Hospital Universitari Mutua de Terrassa, Terrassa, Catalonia